CLINICAL TRIAL: NCT03625414
Title: Comparison of the Physiologic and Biochemical Alterations in the Healthy and Affected Sites of Chronic and Aggressive Periodontitis Patients
Brief Title: Tissue Alterations in Aggressive and Chronic Periodontitis
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hatice Balci Yuce, Dr, Tokat Gaziosmanpasa University
Other Study IDs: balciyuce
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Localized Aggressive Periodontitis; Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gingival biopsies around teeth either affected by periodontal destruction or unaffected. And gingival biopsies of healthy individuals were also obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy individuals: Gingival biopsies of healthy individuals who had no systemic or oral disease or condition.
- Unaffected sites of CP: Chronic periodontitis patients had teeth affected from destruction and some teeth were unaffected. Gingival biopsies of chronic periodontitis patients were taken from sites which were not affected by periodontal destruction.
- Affected sites of CP: Chronic periodontitis patients had teeth affected from destruction and some teeth were unaffected. Gingival biopsies of chronic periodontitis patients were taken from sites which were affected by periodontal destruction.
- Unaffected sites of LAgP: Like chronic periodontitis, aggressive periodontitis patients had also teeth affected by destruction and some teeth were unaffected. Gingival biopsies of aggressive periodontitis patients were taken from sites which were not affected by the periodontal destruction.
- Affected sites of LAgP: Like chronic periodontitis, aggressive periodontitis patients had also teeth affected by destruction and some teeth were unaffected. Gingival biopsies of aggressive periodontitis patients were taken from sites which were affected by the periodontal destruction.

SUMMARY:
Present study intended to compare diseased and healthy sites in chronic and aggressive periodontitis with healthy individuals. The investigators suggest that even unaffected healthy sites of both chronic and aggressive periodontitis patients exhibit subclinical inflammation and tissue destruction with decreased fibroblast cell counts and increased inflammatory cell counts. Investigators also suggest that a possible mechanism which might play a role in the disease progression might occur via a disbalance between matrix metalloproteinases and their inhibitors, and increased hypoxia in diseased sites.

DETAILED DESCRIPTION:
Periodontal disease disrupts soft tissue metabolism in the gingiva through a decrease in the production of collagen, the quality, and quantity of the connective tissue. The etiology and pathogenesis of chronic periodontitis are mostly revealed however, there are many dark points in the etiopathogenesis of aggressive periodontitis. The existence of periodontal destruction at even one tooth in the mouth increases the risk of further periodontal destruction. However, the incidence of progression of the disease to the unaffected teeth was not demonstrated. Yet, the progression of the disease from diseased sites to healthy sites is likely to occur but no evidence is present comparing healthy and diseased sites of chronic and aggressive periodontitis. Present study aimed to evaluate the histological changes in both diseased and healthy sites in both localized aggressive periodontitis (LAgP) and chronic periodontitis (CP) patients by determining fibroblast and inflammatory cell counts in histologic slides and immunohistochemical staining of enzymes and hypoxia markers in order to better understand the dimensions of this demolition in periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

Age range from 30 to 45, the existence of at least 20 functioning teeth, no history of smoking, systemical health, no antibiotic use within 6 months, no periodontal therapy within 6 months, no pregnancy or lactation, no drug use, in addition; For healthy individuals, the existence of oral health

* For localized aggressive periodontitis, the existence of the disease at least for 5 years, the presence of both healthy and diseased sites in the same patient.
* For chronic periodontitis, the existence of the disease at least for 5 years, the presence of both healthy and diseased sites in the same patient.

Exclusion Criteria:

* Patients younger than 30 older than 45 years old, the absence of occlusion, drug use, pregnancy/lactation, smoking, previous antibiotic use, previous periodontal therapy, the existence of any systemical disease.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals, chronic periodontitis patients, and localized aggressive periodontitis patients older than 30 years old and younger than 45 years old were enrolled. The age was specifically chosen because aging changes periodontal and gingival tissues independently of other variables. Any possible factor which might alter connective tissue metabolism were excluded.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Fibroblast and total inflammatory cell counts | Biopsies were obtained a day after initial examinations, histological analysis were performed 2 weeks after.
  Fibroblast and total inflammatory cell counts in the groups were determined in a standardized 1000 micrometer square area with histomorphometric evaluation.

SECONDARY OUTCOMES:
Immunohistochemical staining | Biopsies were obtained a day after initial examinations, histological analysis were performed 2 weeks after
  Expressions of matrix metalloproteinase 8 and tissue inhibitor, hypoxia inducible factor-1alpha and vascular endothelial growth factor were evaluated in histological slides.

CONTACTS AND LOCATIONS:
Overall Officials: HATİCE BALCI YÜCE, PhD, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University Faculty of Dentistry, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No